CLINICAL TRIAL: NCT01109628
Title: Protein Supplementation to Promote Muscle Protein Anabolism in Frail Elderly People
Acronym: ProMuscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Maastricht University Medical Center (Other); Top Institute Food and Nutrition (Other)
Responsible Party: Principal Investigator, Lisette de Groot, Professor, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A1002-1
Record Dates: First submitted 2010-02-12; First posted 2010-04-23 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Sarcopenia
Keywords: sarcopenia; frail elderly; protein drink; skeletal muscle mass; muscle mass in elderly
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protein drink (Experimental)
  Interventions: Dietary Supplement: Protein drink
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Protein drink — Twice a day during 6 months
  Arms: Protein drink
Dietary Supplement: Placebo drink — Twice a day during 6 months
  Arms: Placebo drink

SUMMARY:
The present study is designed to investigate whether timed protein supplementation will increase skeletal muscle mass in the frail elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Frail elderly individuals
* Able to understand and perform the study procedures

Exclusion Criteria:

* Type I or type II diabetes (fasted blood glucose level ≥7,0 mmol)
* No recent history (within 2 years) of participating in any regular resistance exercise training program (general questionnaire)
* Use of anti-coagulation medication (except of Acetyl Salicyl acid)
* Renal insufficiency (eGFR <60 mL/min/1.73 m2)
* Allergic or sensitive for milk proteins

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in skeletal muscle mass | Baseline, 3 months and 6 months

SECONDARY OUTCOMES:
Physical performance | Baseline, 3 months and 6 months
Blood parameters related to the outcome measures | Baseline, 3 months and 6 months
Dietary intake | Baseline, 3 months and 6 months
Physical activity | Baseline, 3 months and 6 months
Cognitive performance | Baseline and 6 months
Blood pressure | Baseline, 3 months and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Derived] van de Rest O, van der Zwaluw NL, Tieland M, Adam JJ, Hiddink GJ, van Loon LJ, de Groot LC. Effect of resistance-type exercise training with or without protein supplementation on cognitive functioning in frail and pre-frail elderly: secondary analysis of a randomized, double-blind, placebo-controlled trial. Mech Ageing Dev. 2014 Mar-Apr;136-137:85-93. doi: 10.1016/j.mad.2013.12.005. Epub 2013 Dec 27. PMID 24374288
- [Derived] van der Zwaluw NL, van de Rest O, Tieland M, Adam JJ, Hiddink GJ, van Loon LJ, de Groot LC. The impact of protein supplementation on cognitive performance in frail elderly. Eur J Nutr. 2014 Apr;53(3):803-12. doi: 10.1007/s00394-013-0584-9. Epub 2013 Sep 18. PMID 24045855
- [Derived] Tieland M, van de Rest O, Dirks ML, van der Zwaluw N, Mensink M, van Loon LJ, de Groot LC. Protein supplementation improves physical performance in frail elderly people: a randomized, double-blind, placebo-controlled trial. J Am Med Dir Assoc. 2012 Oct;13(8):720-6. doi: 10.1016/j.jamda.2012.07.005. Epub 2012 Aug 11. PMID 22889730